CLINICAL TRIAL: NCT00659542
Title: Randomized Study of Mesh Fixation With Absorbable Sutures or Glubran Tissue Sealant in Lichtenstein Hernioplasty
Brief Title: Glubran Mesh Fixation in Lichtenstein Hernioplasty
Acronym: Cyanoacr
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: North Karelia Central Hospital (Other); Paijat-Hame Hospital District (Other)
Responsible Party: Dr. Hannu Paajanen/MD, PhD, Department of Surgery, Kuopio University Hospital, Finland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5204518; cyanoacrylate1
Record Dates: First submitted 2008-04-11; First posted 2008-04-16 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; inguinal hernioplasty; mesh fixation; Lichtenstein hernioplasty
MeSH Terms: conditions — Hernia, Inguinal | interventions — MK 6 cyanoacrylate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): mesh fixation by absorbable sutures
- 2 (Experimental): mesh fixation by cyanoacrylate glue
  Interventions: Procedure: cyanoacrylate glue

INTERVENTIONS:
Procedure: cyanoacrylate glue — 1 ml glue
  Other Names: Glubran2 synthetic surgical glue
  Arms: 2

SUMMARY:
The purpose of the study is to investigate whether chronic postoperative pain is less frequent and quality of life better when inguinal mesh is fixed by using tissue glue compared to conventional sutures in inguinal hernioplasty.

DETAILED DESCRIPTION:
Repair of inguinal hernia in one of the most frequently performed surgical operation in western world. The technique of choice is currently to support inguinal tissues by using polypropylene mesh. Chronic postoperative pain and discomfort occur in 25-30% of patients after inguinal hernioplasty. Pain might be related to mesh fixation by sutures. This randomized study investigates whether mesh fixation by tissue glue (cyanoacrylate) is better than sutures. The patients are followed 1 year postoperatively. Pain, quality of life, operative parameters (time, cost) and recurrences are reported.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia
* adult patient

Exclusion Criteria:

* patient not willing
* multiple recurrences
* inguinal pain without evidence of hernia
* femoral hernia
* large scrotal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 1 year

SECONDARY OUTCOMES:
hernia recurrence, quality of life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Miettinen, MD, PhD, Principal Investigator — University hospital of Kuopio, Finland
Locations (1):
- Hannu Paajanen, Kuopio, Kuopio, Finland

REFERENCES:
- [Background] Ong CC, Jacobsen AS, Joseph VT. Comparing wound closure using tissue glue versus subcuticular suture for pediatric surgical incisions: a prospective, randomised trial. Pediatr Surg Int. 2002 Sep;18(5-6):553-5. doi: 10.1007/s00383-002-0728-0. Epub 2002 Jun 14. PMID 12415411
- [Derived] Matikainen M, Kossi J, Silvasti S, Hulmi T, Paajanen H. Randomized Clinical Trial Comparing Cyanoacrylate Glue Versus Suture Fixation in Lichtenstein Hernia Repair: 7-Year Outcome Analysis. World J Surg. 2017 Jan;41(1):108-113. doi: 10.1007/s00268-016-3801-x. PMID 27864616
- [Derived] Paajanen H, Kossi J, Silvasti S, Hulmi T, Hakala T. Randomized clinical trial of tissue glue versus absorbable sutures for mesh fixation in local anaesthetic Lichtenstein hernia repair. Br J Surg. 2011 Sep;98(9):1245-51. doi: 10.1002/bjs.7598. Epub 2011 Jun 28. PMID 21710480